CLINICAL TRIAL: NCT02994615
Title: Evaluating Microvascular Dysfunction in Symptomatic Patients With HypertroPhic CaRdiomyopathy: The Index of MicrovAscular Resistance (IMR)
Brief Title: Evaluating Microvascular Dysfunction in Symptomatic Patients With HypertroPhic CaRdiomyopathy
Acronym: PRIMARy
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Director of Cardiovascular Interventional Research, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 108627
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Index of Microvascular Resistance; Microvascular dysfunction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypertrophic cardiomyopathy
- Control

SUMMARY:
Patients with hypertrophic cardiomyopathy are being compared to a control group. IMR will be assessed with a pressure wire. Clinical f/u at 3 months and 6 months and a 48 hour holter monitor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Already have an indication for coronary angiography
* Previous diagnosis of hypertrophic cardiomyopathy (unless control)

Exclusion Criteria:

* Fractional flow reserve found to be significant (FFR < 0.8)
* Already have a condition associated with or likely to be associated with an elevated IMR (diabetes, cardiac syndrome X, takotsubo cardiomyopathy, hypertensive cardiomyopathy, severe aortic stenosis, STEMI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic hypertrophic cardiomyopathy versus controls (patients undergoing coronary angiography and FFR
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
IMR in patients with hypertrophic cardiomyopathy (HCM) versus controls | 1 day

SECONDARY OUTCOMES:
Number of ventricular tachycardia | 6 months
  Measured during 48 h recording after 6 months
Chest pain - Canadian Cardiovascular Society (CCS) class | Up to 6 months
Shortness of breath - NYHA class | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, Principal Investigator — London Health Sceinces Centre
Locations (1):
- London Health Sciences Centre, London, Canada

IPD SHARING:
Plan to Share IPD: No